CLINICAL TRIAL: NCT04522180
Title: An Open Label, Randomized, Phase 2 Study to Assess the Safety, Tolerability, and Efficacy of IONIS-GHR-LRx, an Antisense Inhibitor of the Growth Hormone Receptor, Administered Monthly as Monotherapy in Patients With Acromegaly
Brief Title: A Study to Assess the Safety, Tolerability, and Efficacy of IONIS-GHR-LRx Administered in Patients With Acromegaly
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ionis Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ISIS 766720-CS5; 2020-000675-20 (EudraCT Number); NCT04522180 (Other: ClinicalTrials.gov)
Record Dates: First submitted 2020-08-18; First posted 2020-08-21 (Actual); Results first posted 2024-10-03 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-09

CONDITIONS: Acromegaly
Keywords: acromegaly; IONIS-GHR-LRx
MeSH Terms: conditions — Acromegaly

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- GHR-LRX 120 mg (Experimental): Participants received GHR-LRX 120 mg subcutaneous (SC) injection once every month for 73 weeks with a booster dose administered on Day 15 (Week 3).
  Interventions: Drug: GHR-LRX
- GHR-LRX 160 mg (Experimental): Participants received GHR-LRX 160 mg SC injection once every month for 73 weeks with a booster dose administered on Day 15 (Week 3).
  Interventions: Drug: GHR-LRX

INTERVENTIONS:
Drug: GHR-LRX — GHR-LRX was administered by SC injection.
  Other Names: ISIS 766720

SUMMARY:
The purpose of this study was to determine the safety, tolerability, and efficacy of IONIS-GHR-LRx subcutaneous (SC) injection as monotherapy in patients with acromegaly.

DETAILED DESCRIPTION:
This was a multi-center, open-label, randomized, Phase 2 study of IONIS-GHR-LRx in up to 40 participants with acromegaly. Participants were randomized to 1 of 2 treatment groups to receive IONIS GHR-LRx monthly for 73 weeks. At the end of 73 weeks, participants entered a 14-week post-treatment (PT) evaluation period.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females with a documented diagnosis of Acromegaly* who are 18 to 75 years old (inclusive) at the time of informed consent.
2. Have had pituitary surgery (e.g. transsphenoidal) unless there was a contraindication to surgery and are either acromegaly medical treatment naïve, or who had not taken any other acromegaly medications prior to the screening visit as outlined below

   * bromocriptine: 2 weeks
   * cabergoline: 4 weeks
   * quinagolide: 4 weeks
   * octreotide daily injection (SC) or oral formulation: 4 weeks
   * pegvisomant: 4 weeks
   * octreotide LAR: 3 months
   * pasireotide LAR: 4 months
   * lanreotide (all formulations): 3 months
3. At Screening, serum IGF-1 (performed at the central lab) between 1.3 to 5 × ULN, inclusive, adjusted for age and sex.
4. Females must be non-pregnant and non-lactating, and either surgically sterile, post-menopausal, abstinent, or using 1 highly effective method of birth control

Exclusion Criteria:

1. Participants who received surgery for pituitary adenoma within the last 3 months before the trial, and/or planning to receive surgery during the trial
2. Participants who received radiotherapy for pituitary adenoma within the last 2 years before the trial, and/or planning to receive radiotherapy during the trial
3. Participants with a pituitary tumor that, per Investigator judgment, is worsening (e.g., either growing or at risk of compressing or abutting the optic chiasm or other vital structures) as assessed by pituitary/sellar MRI protocol at Screening or within 3 months of Screening. CT scan is allowed if MRI is contraindicated
4. Evidence of decompensated cardiac function per medical judgement and/or New York Heart Association (NYHA) Class 3 or 4
5. Clinical evidence of symptomatic hyperprolactinemia that would necessitate treatment
6. Symptomatic cholelithiasis, and/or choledocholithiasis

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2021-01-04 (Actual); Primary Completion 2022-07-15 (Actual); Study Completion 2023-05-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (22):
- United States (7):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Massachusetts General Hospital, Boston, Massachusetts
  - Palm Research Center Inc., Las Vegas, Nevada
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Cleveland Clinic, Cleveland, Ohio
  - Endocrinology Associates, Inc, Columbus, Ohio
  - Oregon Health & Science University (OHSU), Portland, Oregon
- Estonia (2):
  - East-Tallinn Central Hospital, Tallinn
  - Tartu University Hospital, Tartu
- Debreceni Egyetem Klinikai Kozpont, Debrecen, Hungary
- Italy (2):
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico di Milano, Milan
  - Fondazione Policlinico Universitario A. Gemelli IRCCS - Universita Cattolica del Sacro Cuore, Roma
- Pauls Stradins Clinical University Hospital, Riga, Latvia
- Lithuania (2):
  - Vaidoto Urbanaviciaus Individuali imone, Alytus
  - Hospital of Lithuanian University of Health Sciences (LSMU) Kauno klinikos, Kaunas
- Poland (3):
  - Zespol Oddzialow Chorob Wewnetrznych, Endokrynologii i Diabetologii, Warsaw
  - Uniwersytecki Szpital Kliniczny, im. Jana Mikulicza-Radeckiego we Wroclawiu,, Wroclaw
  - Centrum Badan Klinicznych Piotr Napora Lekarze Sp. p., Wroclaw
- Centrul Medical Unirea Bucuresti, Endocrinologie, Bucharest, Romania
- I.M. Sechenov Moscow First State Medical University, Moscow, Russia
- Serbia (2):
  - Clinical Center of Serbia, Belgrade
  - Clinical Center of Vojvodina, Novi Sad

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 22 investigational sites in United States of America, Estonia, Hungary, Italy, Latvia, Lithuania, Poland, Romania, Russia, and Serbia from 4 January 2021 to 18Jan2022.
Pre-assignment Details: Participants with acromegaly were enrolled and assigned to receive an initial dose of GHR-LRX 120 mg or GHR-LRX 160 mg up to week 17 (when the first post-baseline IGF-1 results were available). After Week 17, patients may have received a higher dose up to 160 mg for efficacy, if necessary, up to 73 weeks.
Period: Overall Study
Arm/Group | GHR-LRX 120 mg | GHR-LRX 160 mg
Started | 18 | 16
Per Protocol Set (Initial Dose) (Per protocol set included all participants that started the study and who completed at least 6 of the 8 doses of GHR-LRX with the first 27 Weeks administered and had no significant protocol deviations that impacted efficacy. Initial dose was the dose received up to Week 17 and maximum dose was the dose received following dose escalation up to Week 73.) | 18 | 14
Increased Dose From Initial 120mg to Maximum Dose 160mg (Week 17 to Week 45) | 15 | 0
Completed (Completed included participants who completed the study treatment.) | 5 | 3
Not Completed | 13 | 13
Not completed — Investigator judgement | 3 | 4
Not completed — Voluntary withdrawal | 1 | 0
Not completed — Pregnancy | 0 | 1
Not completed — Adverse Event or Serious Adverse event | 1 | 3
Not completed — Reason not specified | 8 | 5

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all participants who were randomized and received at least 1 dose of GHR-LRX
Groups:
- Total: Total of all reporting groups
Arm/Group | GHR-LRX 120 mg | GHR-LRX 160 mg | Total
Number analyzed (Participants) | 3 | 31 | 34
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.0 (3.46) | 51.9 (11.76) | 52.9 (11.68)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 16 | 17
  Male | 2 | 15 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 31 | 34
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 3 | 30 | 33
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Insulin-like Growth Factor I (IGF-1) From Baseline to Week 27
Description: IGF-1 is a hormone that manages the effects of growth hormone (GH) in the body. Baseline of IGF-1 is defined as the average value of Screening and Day 1. A negative percent change from Baseline indicated improvement.
Time Frame: Baseline to Week 27
Population: Per protocol set (total dose) included all FAS participants who completed at least 6 of the 8 doses of GHR-LRX with the first 27 Weeks administered and have no significant protocol deviations that would be expected to impact efficacy. Total dose includes results for IGF-1 reduction that combines both 120 mg and 160 mg doses. Analysis based on highest dose received as prespecified in the statistical analysis plan (SAP).
Measure: Mean (Standard Deviation); unit: Percent change
Groups:
- GHR-LRX 120 mg (Per Protocol Set): Participants received a maximum dose of GHR-LRX 120 mg SC injection once every month for up to 73 weeks with a booster dose administered on Day 15 (Week 3).
- GHR-LRX 160 mg (Per Protocol Set): Participants received a maximum dose of GHR-LRX 160 mg SC injection once every month for up to 73 weeks with a booster dose administered on Day 15 (Week 3).
- GHR-LRX Total (Per Protocol Set): Overall number of participants analyzed is the number of participants available for analyses. Total of all participants in the Per Protocol Set (received maximum doses of 120 mg or 160 mg doses).
Arm/Group | GHR-LRX 120 mg (Per Protocol Set) | GHR-LRX 160 mg (Per Protocol Set) | GHR-LRX Total (Per Protocol Set)
Number analyzed (Participants) | 2 | 24 | 26
Percent change | -6.20 (10.803) | -7.16 (20.100) | -7.09 (19.402)

2. Secondary Outcome: Percentage of Participants Who Achieve Normalized IGF-1 Levels to Within 1.2 Times Gender and Age Limits at Day 183 (Week 27)
Description: Normalized IGF-1 level is defined as the ratio of the serum IGF-1 level and the participant's upper limit of normal (ULN).
Time Frame: At Week 27
Population: Per protocol set (initial dose) includes all FAS participants who completed at least 6 of the 8 doses of GHR-LRX within the first 27 weeks administered and had no significant protocol deviations that would have been expected to impact efficacy. Here, overall number of participants analyzed signifies the number of participants available for analyses. Analysis based on highest dose received as prespecified in the statistical analysis plan (SAP).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- GHR-LRX 120 mg: Participants received a maximum dose of GHR-LRX 120 mg SC injection once every month for up to 73 weeks with a booster dose administered on Day 15 (Week 3).
- GHR-LRX 160 mg: Participants received a maximum dose of GHR-LRX 160 mg SC injection once every month for up to 73 weeks with a booster dose administered on Day 15 (Week 3).
- GHR-LRX Total: Overall number of participants analyzed is the number of participants available for analyses. Total of all participants in the Per Protocol Set (received maximum doses of 120 mg or 160 mg doses).
Arm/Group | GHR-LRX 120 mg | GHR-LRX 160 mg | GHR-LRX Total
Number analyzed (Participants) | 2 | 24 | 26
percentage of participants | 0 [0.0 to 84.2] | 0 [0.0 to 14.2] | 0 [0.0 to 13.2]

3. Secondary Outcome: Percentage of Participants Who Achieve Normalized IGF-1 Levels to Within 1.0 Times Gender and Age Limits at Day 183 (Week 27)
Description: Normalized IGF-1 level is defined as the ratio of the serum IGF-1 level and the participant's ULN.
Time Frame: At Week 27
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | GHR-LRX 120 mg | GHR-LRX 160 mg | GHR-LRX Total
Number analyzed (Participants) | 2 | 24 | 26
percentage of participants | 0 [0.0 to 84.2] | 0 [0.0 to 14.2] | 0 [0.0 to 13.2]

4. Secondary Outcome: Change From Baseline in Serum IGF-1 Over Time
Description: IGF-1 is a hormone that manages the effects of growth hormone (GH) in the body. A negative change from baseline indicated improvement.
Time Frame: Up to approximately 80 weeks
Population: Per protocol set (maximum dose) includes all FAS participants who completed at least 6 of the 8 doses of GHR-LRX within the first 27 weeks administered and had no significant protocol deviations that would have been expected to impact efficacy. Here, 'Number analyzed' signifies the number of participants analyzed at specified time points.
Measure: Mean (Standard Deviation); unit: nanograms per milliliter (ng/mL)
Groups:
- GHR-LRX 120 mg: Participants received maximum dose of GHR-LRX 120 mg SC injection once every month for up to 73 weeks with a booster dose administered on Day 15 (Week 3).
- GHR-LRX 160 mg: Participants received maximum dose of GHR-LRX 160 mg SC injection once every month for up to 73 weeks with a booster dose administered on Day 15 (Week 3).
Arm/Group | GHR-LRX 120 mg | GHR-LRX 160 mg | GHR-LRX Total
Number analyzed (Participants) | 3 | 29 | 32
nanograms per milliliter (ng/mL)
  At Week 3 | -30.00 (44.908) | 5.03 (49.932) | 1.74 (49.896)
  At Week 5 | -50.67 (101.186) | -45.53 (87.817) | -46.01 (87.341)
  Week 7 | -84.33 (133.829) | -39.46 (80.258) | -43.66 (84.558)
  Week 9 | -109.00 (111.959) | -25.28 (93.924) | -33.13 (96.909)
  Week 11 | -157.67 (144.923) | -14.28 (64.463) | -27.73 (83.134)
  Week 13 | -89.67 (130.989) | -38.01 (68.885) | -42.85 (75.013)
  Week 15: number analyzed (Participants) | 3 | 27 | 30
  Week 15 | -112.00 (112.618) | -28.97 (79.942) | -37.28 (85.124)
  Week 17 | -89.33 (136.433) | 136.433 (88.212) | -41.82 (92.034)
  Week 21: number analyzed (Participants) | 2 | 24 | 26
  Week 21 | -123.25 (136.118) | -51.91 (92.746) | -57.39 (95.030)
  Week 25: number analyzed (Participants) | 2 | 24 | 26
  Week 25 | -99.75 (126.926) | -36.99 (78.236) | -41.82 (81.034)
  Week 27: number analyzed (Participants) | 2 | 24 | 26
  Week 27 | -58.75 (87.328) | -49.45 (112.579) | -50.16 (109.415)
  Week 29: number analyzed (Participants) | 2 | 23 | 25
  Week 29 | -90.25 (126.219) | -40.25 (80.174) | -44.25 (82.145)
  Week 33: number analyzed (Participants) | 2 | 23 | 25
  Week 33 | -75.25 (110.662) | -53.12 (72.494) | -54.89 (73.247)
  Week 37: number analyzed (Participants) | 2 | 23 | 25
  Week 37 | -98.75 (179.252) | -32.55 (107.499) | -37.85 (110.760)
  Week 41: number analyzed (Participants) | 2 | 23 | 25
  Week 41 | -93.25 (146.018) | -43.12 (97.911) | -47.13 (99.341)
  Week 45: number analyzed (Participants) | 2 | 21 | 23
  Week 45 | -86.75 (175.009) | -52.80 (110.595) | -55.75 (112.282)
  Week 49: number analyzed (Participants) | 2 | 19 | 21
  Week 49 | -81.75 (109.955) | -64.59 (105.493) | -66.23 (103.184)
  Week 53: number analyzed (Participants) | 2 | 18 | 20
  Week 53 | -90.25 (158.745) | -68.71 (81.822) | -70.86 (85.793)
  Week 57: number analyzed (Participants) | 2 | 17 | 19
  Week 57 | -73.75 (91.570) | -59.43 (90.080) | -60.93 (87.744)
  Week 61: number analyzed (Participants) | 2 | 15 | 17
  Week 61 | -125.75 (199.051) | -83.08 (112.428) | -88.10 (117.206)
  Week 65: number analyzed (Participants) | 1 | 11 | 12
  Week 65 | 74.00 (NA) — Due to one participant, standard deviation (SD) was not estimable. | -103.30 (102.760) | -88.52 (110.540)
  Week 69: number analyzed (Participants) | 1 | 8 | 9
  Week 69 | -22.00 (NA) — Due to one participant, standard deviation (SD) was not estimable. | -85.59 (53.018) | -78.53 (53.934)
  Week 73: number analyzed (Participants) | 1 | 7 | 8
  Week 73 | -1.00 (NA) — Due to one participant, standard deviation (SD) was not estimable. | -91.18 (79.166) | -79.91 (79.928)

5. Secondary Outcome: Percent Change From Baseline in Serum IGF-1 Over Time
Description: IGF-1 is a hormone that manages the effects of growth hormone (GH) in the body. A negative percent change from Baseline indicated improvement.
Time Frame: Baseline, Week 3, 5, 7, 9, 11, 13, 15, 17, 21, 25, 27, 29, 33, 37, 41, 45, 49, 53, 57, 61, 65, 69, 73
Population: Per protocol set (maximum dose) includes all FAS participants who completed at least 6 of the 8 doses of GHR-LRX within the first 27 weeks administered and had no significant protocol deviations that would have been expected to impact efficacy. 'Number analyzed' signifies the number of participants analyzed at specified time points.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | GHR-LRX 120 mg | GHR-LRX 160 mg | GHR-LRX Total
Number analyzed (Participants) | 3 | 29 | 32
percent change
  At Week 3 | -3.73 (5.072) | 2.64 (11.936) | 2.04 (11.571)
  At Week 5 | -5.67 (12.296) | -8.28 (18.158) | -8.04 (17.554)
  At Week 7 | -9.57 (16.297) | -7.16 (16.637) | -7.39 (16.360)
  At Week 9 | -17.43 (11.285) | -2.95 (16.995) | -4.31 (16.955)
  At Week 11 | -26.56 (15.966) | -1.15 (16.235) | -3.54 (17.638)
  At Week 13 | -10.32 (17.934) | -6.35 (16.837) | -6.72 (16.679)
  At Week 15: number analyzed (Participants) | 3 | 27 | 30
  At Week 15 | -17.81 (13.377) | -5.40 (21.168) | -6.64 (20.698)
  At Week 17 | -9.36 (20.529) | -4.59 (20.631) | -5.04 (20.338)
  At Week 21: number analyzed (Participants) | 2 | 24 | 26
  At Week 21 | -19.07 (8.695) | -9.98 (22.994) | -10.68 (22.261)
  At Week 25: number analyzed (Participants) | 2 | 24 | 26
  At Week 25 | -13.28 (12.010) | -6.58 (16.164) | -7.10 (15.794)
  At Week 27: number analyzed (Participants) | 2 | 24 | 26
  At Week 27 | -6.20 (10.803) | -7.16 (20.100) | -7.09 (19.402)
  At Week 29: number analyzed (Participants) | 2 | 23 | 25
  At Week 29 | -10.55 (14.242) | -7.92 (18.173) | -8.13 (17.656)
  At Week 33: number analyzed (Participants) | 2 | 23 | 25
  At Week 33 | -8.10 (13.484) | -10.10 (16.351) | -9.94 (15.905)
  At Week 37: number analyzed (Participants) | 2 | 23 | 25
  At Week 37 | -6.25 (27.791) | -4.29 (25.161) | -4.45 (24.755)
  At Week 41: number analyzed (Participants) | 2 | 23 | 25
  At Week 41 | -8.89 (19.345) | -9.01 (23.250) | -9.00 (22.608)
  At Week 45: number analyzed (Participants) | 2 | 21 | 23
  At Week 45 | -3.24 (29.617) | -8.26 (23.791) | -7.82 (23.590)
  At Week 49: number analyzed (Participants) | 2 | 19 | 21
  At Week 49 | -10.12 (11.603) | -12.83 (22.932) | -12.57 (21.924)
  At Week 53: number analyzed (Participants) | 2 | 18 | 20
  At Week 53 | -6.37 (23.892) | -14.81 (19.811) | -13.97 (19.697)
  At Week 57: number analyzed (Participants) | 2 | 17 | 19
  At Week 57 | -10.11 (8.205) | -10.50 (19.795) | -10.46 (18.763)
  At Week 61: number analyzed (Participants) | 2 | 15 | 17
  At Week 61 | -11.72 (26.723) | -18.94 (25.675) | -18.09 (25.044)
  At Week 65: number analyzed (Participants) | 1 | 11 | 12
  At Week 65 | 35.41 (NA) — Due to one participant, standard deviation (SD) was not estimable. | -21.36 (25.392) | -16.63 (29.235)
  At Week 69: number analyzed (Participants) | 1 | 8 | 9
  At Week 69 | -10.53 (NA) — Due to one participant, standard deviation (SD) was not estimable. | -23.32 (14.391) | -21.89 (14.120)
  At Week 73: number analyzed (Participants) | 1 | 7 | 8
  At Week 73 | -0.48 (NA) — Due to one participant, standard deviation (SD) was not estimable. | -22.62 (20.556) | -19.85 (20.578)

ADVERSE EVENTS:
Time Frame: From Day 1 up to the end of study follow-up (up to week 121).
Description: All participants who were randomized and received at least 1 dose of GHR-LRX. Data for all-cause mortality, serious and non-serious adverse events is reported as per the maximum dose received by participants per arm considering dose escalation was allowed in this study. Adverse events collected based on highest dose received as prespecified in the statistical analysis plan (SAP).
Groups:
- GHR-LRX 120 mg (Safety Set): Participants received a maximum dose of GHR-LRX 120 mg SC injection once every month for up to 73 weeks with a booster dose administered on Day 15 (Week 3).
- GHR-LRX 160 mg (Safety Set): Participants received a maximum dose of GHR-LRX 160 mg SC injection once every month for up to 73 weeks with a booster dose administered on Day 15 (Week 3). Due to the length of the study after Week 17, participants received the maximum dose longer than the initial dose.
- GHR-LRX Total (Safety Set): Overall number of participants (34) analyzed is the number of participants available for analyses.
Arm/Group | GHR-LRX 120 mg (Safety Set) | GHR-LRX 160 mg (Safety Set) | GHR-LRX Total (Safety Set)
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/31 | 0/34
Serious Adverse Events (participants affected / at risk) | 1/3 | 2/31 | 3/34
Other Adverse Events (participants affected / at risk) | 3/3 | 26/31 | 29/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GHR-LRX 120 mg (Safety Set) (N=3) | GHR-LRX 160 mg (Safety Set) (N=31) | GHR-LRX Total (Safety Set) (N=34)
Atrioventricular block second degree (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
COVID-19 pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Cholecystitis chronic (Hepatobiliary disorders) | 0 (0) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | GHR-LRX 120 mg (Safety Set) (N=3) | GHR-LRX 160 mg (Safety Set) (N=31) | GHR-LRX Total (Safety Set) (N=34)
COVID-19 (Infections and infestations) | 1 | 6 | 7
Respiratory tract infection viral (Infections and infestations) | 1 | 3 | 4
Urinary tract infection (Infections and infestations) | 0 | 4 | 4
Nasopharyngitis (Infections and infestations) | 0 | 3 | 3
Asymptomatic COVID-19 (Infections and infestations) | 0 | 2 | 2
Respiratory tract infection (Infections and infestations) | 0 | 2 | 2
Rhinitis (Infections and infestations) | 0 | 2 | 2
Upper respiratory tract infection (Infections and infestations) | 0 | 2 | 2
Pyelonephritis chronic (Infections and infestations) | 1 | 0 | 1
Headache (Nervous system disorders) | 0 | 11 | 11
Dizziness (Nervous system disorders) | 0 | 3 | 3
Dysgeusia (Nervous system disorders) | 0 | 2 | 2
Paraesthesia (Nervous system disorders) | 0 | 2 | 2
Tremor (Nervous system disorders) | 1 | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 4 | 5
Dyspepsia (Gastrointestinal disorders) | 0 | 4 | 4
Diarrhoea (Gastrointestinal disorders) | 0 | 3 | 3
Abdominal pain (Gastrointestinal disorders) | 0 | 2 | 2
Diverticulum intestinal (Gastrointestinal disorders) | 0 | 2 | 2
Flatulence (Gastrointestinal disorders) | 1 | 1 | 2
Haematochezia (Gastrointestinal disorders) | 0 | 2 | 2
Haemorrhoids (Gastrointestinal disorders) | 1 | 1 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 3 | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 2 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 2
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Blood creatine phosphokinase increased (Investigations) | 0 | 3 | 3
Lipase increased (Investigations) | 0 | 2 | 2
Urine albumin/creatinine ratio increased (Investigations) | 0 | 2 | 2
Weight increased (Investigations) | 0 | 2 | 2
Asthenia (General disorders) | 1 | 4 | 5
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 2 | 2
Rash (Skin and subcutaneous tissue disorders) | 0 | 2 | 2
Dermal cyst (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Rosacea (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Hypertension (Vascular disorders) | 0 | 5 | 5
Dyslipidaemia (Metabolism and nutrition disorders) | 0 | 2 | 2
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 | 1 | 2
Anaemia (Blood and lymphatic system disorders) | 1 | 2 | 3
Sinus bradycardia (Cardiac disorders) | 0 | 3 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 2
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 2 | 2
Vision blurred (Eye disorders) | 0 | 2 | 2
Insomnia (Psychiatric disorders) | 0 | 2 | 2
Renal cyst (Renal and urinary disorders) | 2 | 0 | 2
Hepatic cyst (Hepatobiliary disorders) | 1 | 0 | 1
Hepatic steatosis (Hepatobiliary disorders) | 1 | 0 | 1
Post procedural hypothyroidism (Injury, poisoning and procedural complications) | 1 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Principal investigators are not employees of Ionis Pharmaceuticals. Work with CDT to establish the Principal Investigator agreement.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-08-30): https://cdn.clinicaltrials.gov/large-docs/80/NCT04522180/Prot_SAP_000.pdf